CLINICAL TRIAL: NCT05161052
Title: Assessment of Corneal Stiffness Parameters in Keratoconus After Corneal Collagen Cross Linking Using Dynamic Scheimpflug Technology and Anterior Segment Optical Coherence Tomography.
Brief Title: Assessment of Corneal Stiffness in Keratoconus After Crosslinking by Corvis ST and OCT.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Mohamed Samir Elnoamany, Principal Investigator, Cairo University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MD-80-2021
Record Dates: First submitted 2021-10-19; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Intervention Model Description: * Measurement of corneal stiffness parameters { Deformation Amplitude (DAR1), Integrated radius, Stress parameter (SP A1), Stress strain index (SSI) and Corvis biomechanical index (CBI) } in keratoconic corneas before and after 3 and 6 months CXL using Corvis ST.
  * Measurement of demarcation line depth using anterior segment OCT and correlate between corneal stiffness following CXL and demarcation line depth.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Corvis ST (dynamic Scheimpflug technology) — * Measurement of corneal stiffness parameters { Deformation Amlitude (DAR1), Integrated radius, Stress parameter (SP A1), Stress strain index (SSI) and Corvis biomechanical index (CBI) } in keratoconic corneas before and after 3 and 6 months CXL using Corvis ST.
  * Measurement of demarcation line depth using anterior segment OCT and correlate between corneal stiffness following CXL and demarcation line depth
  Other Names: OCT (Optical Coherence tomography)

SUMMARY:
Objectives:

* Measurement of corneal stiffness parameters { Deformation Amlitude (DAR1), Integrated radius, Stress parameter (SP A1), Stress strain index (SSI) and Corvis biomechanical index (CBI) } in keratoconic corneas before and after 3 and 6 months CXL using Corvis ST.
* Measurement of demarcation line depth using anterior segment OCT and correlate between corneal stiffness following CXL and demarcation line depth.

DETAILED DESCRIPTION:
Background and Rationale:

Keratoconus is a progressive corneal degeneration resulting from noninflammatory thinning of the corneal stroma. Visual impairment typically commences in adolescence and progresses thereafter. Further increase in myopia, irregular astigmatism, and subepithelial scarring leads to visual impairment. Treatment modalities are based on refractive correction with spectacles or contact lenses to correct astigmatism and restore visual acuity. Such modalities do not stop ectatic progression and further visual deterioration, which ultimately necessitates corneal transplantation in 10% to 20% of patients.

Corneal collagen cross-linking (CXL) has emerged as a promising techniq;ue to slow or halt the progression of keratoconus. CXL leads to an increase in intra and interfibrillar covalent bonds by photosensitized oxidation and causes a biomechanical stabilization of the cornea.

Corneal visualization using dynamic Scheimpflug technology (Corvis ST, Oculus Optikger€ate GmbH) allows in vivo measurement of the corneal biomechanical deformation response to an applied air puff and is useful for evaluating the biomechanical response parameters of the cornea. It captures the dynamic corneal deformation caused by an air puff using an ultrahigh- speed camera that operates at a speed of greater than 4300 frames per second to capture a series of 140 sequential horizontal Scheimpflug images of the temporal-nasal cross section of the cornea. The consistency of the air puff has been shown and the spatial and temporal profiles have been characterized to allow calculation of the load on the cornea within the imaging window.

The Corvis ST enables the measurement of several parameters by analyzing the timing and patterns of deformation at the highest concavity as well as applanation during inward deformation (loading) and outward recovery (unloading). The original parameters have been reported to be influenced most strongly by intraocular pressure (IOP) as well as age and central corneal thickness (CCT). Recently, new corneal biomechanical parameters were introduced, including the Deformation Amplitude ratio at 1.0 mm (DAR1), Deformation Amplitude ratio at 2.0 mm (DAR2), Integrated radius, Stiffness Parameter at first applanation (SP A1), Ambrosio's Relational Thickness (ARTH) , Corbic Biomechanical index (CBI) and biomechanically corrected IOP (bIOP).

Laboratory studies have shown that the effective depth of CXL is confined to the anterior 300 μm of the cornea. Moreover, a stromal demarcation line between treated and untreated stroma was visible biomicroscopically at a depth of approximately 300 μm over the entire cornea after CXL treatment. This demarcation line was also evident on optical coherence tomography (OCT). The depth of this line has been postulated as an indirect measurement of cross-linking effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented progressive keratoconus within one year include any of the following:

A. ≥ 1.00 diopter increase in maximal keratometry (Kmax). B. ≥ 1.00 diopter increase in the manifest cylinder. C. ≥ 0.75 diopter increase in average of Kmax and Kmin (Kmean). D. ≥ 2% decrease in central thickness. E. ≥ 1.50 diopter increase in the central K power from baseline. F. ≥ 1.0 diopter increase in manifest spherical equivalent change (MRSE).

* All patients have minimal corneal stromal thickness 400 μm before UVA irradiation.

Exclusion Criteria:

* Patients with corneal rings.
* Advanced keratoconus with corneal scarring.
* History of herpetic keratitis and severe corneal infection.
* Pregnancy or breastfeeding.
* The use of rigid contact lens¬es for more than 4 weeks before the baseline evaluation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Patients between 18- 40 years old with progressive keratoconus undergoing CXL.
Enrollment: 55 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Measuring changes in corneal stiffness parameters in keratoconus after CXL by Corvis ST which measures corneal stiffness parameters. | Before crosslinknig procedure and after 3, 6 months using Corvis ST.
  Measurement of changes in corneal stiffness parameters { Deformation Amplitude (DAR1), Integrated radius, Stress parameter (SP A1), Stress strain index (SSI) and Corvis biomechanical index (CBI) } before and after crosslinking procedure to measure corneal stiffness.

OTHER OUTCOMES:
Measuring demarcation line depth in microns by anterior segment OCT. in keratoconus after CXL with demarcation line depth in microns by anterior segment OCT. | After 3 and 6 months using anterior segment OCT
  Measurement of demarcation line depth in the cornea in microns using anterior segment OCT which gives an indicator to corneal stiffness after crosslinking procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Fakhry, MD, Principal Investigator — Cairo University

REFERENCES:
- [Background] Salouti R, Bagheri M, Shamsi A, Zamani M. Corneal Parameters in Healthy Subjects Assessed by Corvis ST. J Ophthalmic Vis Res. 2020 Feb 2;15(1):24-31. doi: 10.18502/jovr.v15i1.5936. eCollection 2020 Jan-Mar. PMID 32095205
- [Background] Nakao Y, Kiuchi Y, Okumichi H. Evaluation of biomechanically corrected intraocular pressure using Corvis ST and comparison of the Corvis ST, noncontact tonometer, and Goldmann applanation tonometer in patients with glaucoma. PLoS One. 2020 Sep 23;15(9):e0238395. doi: 10.1371/journal.pone.0238395. eCollection 2020. PMID 32966284
- [Background] Herber R, Terai N, Pillunat KR, Raiskup F, Pillunat LE, Sporl E. [Dynamic Scheimpflug Analyzer (Corvis ST) for measurement of corneal biomechanical parameters : A praxis-related overview]. Ophthalmologe. 2018 Aug;115(8):635-643. doi: 10.1007/s00347-018-0716-y. German. PMID 29767348